CLINICAL TRIAL: NCT06069570
Title: Phase 1 Trial Evaluating the Safety and Tolerability of Gamma Delta T-Cell Infusions in Combination With Low Dose Radiotherapy in Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer or Solid Tumors With Bone Metastases
Brief Title: Safety Study for a Gamma Delta T Cell Product Used With Low Dose Radiotherapy in Patients With Locally Advanced or Metastatic NSCLC or Solid Tumors With Bone Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kiromic BioPharma Inc. (Industry)
Collaborators: Stiris Research Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DELTACEL-01
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung Cancer; Bone Metastases From Solid Tumors
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: The maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) or the maximum administered dose (MAD) will be determined based on isotonic regression in Part 1 Dose Escalation. If the MTD/MAD shows an acceptable safety and tolerability profile, an additional 12 participants in Part 2 expansion will be enrolled. Three dose levels of KB-GDT-01 will be evaluated and will follow a Bayesian Optimal Interval (BOIN) design rule based on a targeting rate of 25% for dose limiting toxicity (DLT) occurring between the first KB-GDT-01 infusion and Day 40. Depending on observed DLT rate, the safety monitoring committee will assess whether to escalate to the next dose, de-escalate (not applicable for the first dose), hold at current dose or stop the study if at the first dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- KB-GDT-01 cells (Experimental): Dose Level 1: 400 x10^6, 800 x10^6 or 1600 x10^6 KB-GDT-01 cells + radiation (1.0 Gy/fraction)
  Interventions: Biological: KB-GDT-01

INTERVENTIONS:
Biological: KB-GDT-01 — KB-GDT-01 is an allogeneic, gamma delta T-cell suspension product manufactured from the isolation of healthy donor peripheral blood mononuclear cells (PBMC). The KB-GDT-01 cells are cryopreserved in vapor phase liquid nitrogen (LN2) in 50 mL CryoMACS® cryobags for a total of 200 × 106 viable cells/bag. The KB-GDT-01 cryopreserved product is thawed and administered intravenously (IV) until the entire bag is infused by gravity. Low dose radiotherapy (LDRT) will be administered to selected tumor sites (maximum of 5 isocenters) at 1.0 Gy/fraction on Days 1 and 2, followed by the KB-GDT-01 IV infusion on Day 3. LDRT will be repeated on Days 8 and 9, and the 2nd KB-GDT-01 IV infusion on Day 10.
  Other Names: Low dose radiotherapy

SUMMARY:
This is a clinical trial studying intravenous infusions of allogeneic gamma delta T cells after receiving low dose radiotherapy in participants with locally advanced or metastatic non-small cell lung cancer or solid tumors with bone metastases to evaluate the safety and efficacy of combining immunotherapy with radiation therapy.

DETAILED DESCRIPTION:
In this clinical trial, or 'study', participants with locally advanced or metastatic, non-small cell cancer (NSCLC) or solid tumors with bone metastases, will receive KB-GDT-01, an allogeneic (cells from healthy donors) gamma delta T-cell product. All participants will receive KB-GDT-01 as intravenous infusions in combination with radiotherapy.

After being informed about the study and its potential risks, during the 28-day screening period, all consented participants will have laboratory tests, assessments, tumor scans, and a tumor biopsy.

Cytokine release syndrome symptoms and other potential adverse effects, will be monitored during the dose limiting toxicity period.

The study will be conducted in 2 parts, with the same number of visits in each part.

In Part 1 Dose Escalation, the study will attempt to identify the best dose with the lowest incidence of adverse effects (AE) and try to identify if the KB-GDT-01 is working (effectiveness). In Part 2 Dose Expansion the best dose will be further investigated for AE and effectiveness. There will be up to 36 participants in Part 1 and up to 21 additional participants in Part 2 of the study.

The total treatment period of the study drug protocol will be completed in 31 days. Participants will then attend clinic visits during a 30-day short-term follow-up period, with a subsequent long-term follow-up period up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form.
* Male or female, > 18 years old.
* Minimum body weight of 50 kilograms (kg).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Histologically or cytologically confirmed locally advanced or metastatic NSCLC or locally advanced or metastatic solid tumor with bone metastasis
* Progressed on SOC therapy including platinum-based chemotherapy and immune checkpoint inhibitors (NSCLC), and are not a candidate for further standard anti-neoplastic therapy and/or have exhibited intolerance to and/or declined clinically applicable salvage therapies, and/or have declined therapy.
* Genomic screening, with tumors with known actionable molecular alterations, such as EGFR, ALK, ROS-1, BRAF, RET, MET, and KRAS etc., must have progressed on appropriate target-directed molecular therapy.
* At least one measurable target lesion based on RECIST v1.1 confirmed by radiological imaging. Participants with isolated bone metastases are eligible for enrollment are not required to have measurable disease
* All toxicity associated with previous treatments are recovered to CTCAE grade of ≤1, except for continuing alopecia.
* Adequate hematopoietic, hepatic and renal function
* Agree to adequate contraception for up to 120 days after the last dose of study drug.
* Negative serum pregnancy test for women of childbearing potential
* All primary and metastatic disease sites are amenable to LDRT
* For solid tumors with bone metastases subjects (Part 2 Cohort B): receiving zoledronic acid for solid tumors with bone metastases

Exclusion Criteria:

* Chemotherapy, investigational, and/or check-point inhibitor therapy within the 30 days prior to study Day 1.
* Major surgery, except for vascular access placement, within the 30 days prior to study Day 1.
* Active autoimmune disease requiring immunosuppressive therapy.
* Infection requiring systemic treatment within 30 days prior to study Day 1.
* History of peritoneal effusion (ascites), pericardial, or pleural effusions/nodules.
* Uncontrolled hypertension, history of arrhythmia including atrial fibrillation, unstable angina, decompensated congestive heart failure, cardiac ejection fraction ≤ 50%, myocardial infarction, or marked baseline prolonged QT/QTc intervals.
* Human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C detection.
* Participation in the treatment portion of a clinical trial or completed a clinical trial within the 30 days prior to the first dose of KB-GDT-01.
* Presence of any condition that may, in the opinion of the Investigator, render the patient inappropriate from participating in the study.
* Breastfeeding or pregnant female, or patient is expecting to conceive or father children during the study.
* Allergy or intolerance to any of the study product ingredients or excipients.
* Live vaccines administered within 30 days prior to study Day 1.
* Individuals lacking capacity to consent for themselves.
* Superior vena cava obstruction
* Prior radiation therapy to a selected LDRT treatment site </= 30 days prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AE) and/or Dose Limiting Toxicities (DLT) as a Measurement of Safety and Tolerability of KB-GDT-01 in Combination with LDRT | From the first infusion of study drug until Day 40 or 30 days after the last study drug infusion, whichever occurs later
  DLT, defined as the occurrence or start of a clinically significant Grade 3 or greater AE (per CTCAE v5.0) occurring during the DLT assessment period that cannot be attributed to disease progression, intercurrent illness, or concomitant medication.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From first study drug infusion through to Month 24
  Investigator assessed ORR per RECIST v1.1. ORR is defined as the percentage of participants with a best overall response of complete or partial response.
Progression Free Survival (PFS) | From first study drug infusion until the first evidence of disease progression, death or Month 24.
  Investigator assessed PFS per RECIST v1.1. PFS is defined as the time from first study drug infusion until the first evidence of disease progression or death.
Overall Survival (OS) | From first study drug infusion until death or Month 24.
  Investigator assessed OS per RECIST v1.1. OS is defined as the time from first study drug infusion to death.
Time to Progression (TTP) | From first study drug infusion until first evidence of disease progression or Month 24.
  Investigator assessed TTP per RECIST v1.1. TTP is defined as the time from first study drug infusion until first evidence of disease progression.
Time to Treatment Response (TTR) | From first study drug infusion until first evidence of disease response or Month 24.
  Investigator assessed TTR per RECIST v1.1. TTR is defined as the time from first study drug infusion until first evidence of disease response.
Disease Control Rate (DCR) | From first study drug infusion until first evidence of disease response or stable disease or Month 24.
  Investigator assessed DCR per RECIST v1.1 DCR is defined as the percentage of participants with complete response, partial response or stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Luke, MD, FACP, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia